CLINICAL TRIAL: NCT04393233
Title: Drug Management of Rheumatoid Arthritis in Covid-19 Context : Impact on Therapeutic De-escalation
Acronym: RHUMACOVID
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RHUMACOVID ( 29BRC20.0110)
Record Dates: First submitted 2020-04-22; First posted 2020-05-19 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2020-04

CONDITIONS: Rheumatoid Arthritis; COVID
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current situation of Sars-Cov-2 pandemic generates fears in the general population. Among patients receiving long-term immunomodulatory drugs, especially in the context of auto-immune diseases, there may be legitimates interrogations about the appropriateness of continuing treatment, without modification, in the current context. Most patients with Juvenile Rheumatoid Arthritis benefit from long-term immunmodulatory therapy (DMARD - disease modifying anti-rheumatic drug), more or less combined with regular use of non-steroidal anti-inflammatory drugs (NSAIDs) or corticosteroids.The present study will characterize this issue by defining the proportion of patients whose usual treatment of Rheumatoid Arthritis has been modified in relation to the actual sanitary crisis.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis satisfying ACR/EULAR criteria
* Ongoing DMARD therapy

Exclusion Criteria:

* Inhability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients with ongoing DMARD therapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-08-23 (Actual); Study Completion 2020-08-23 (Actual)

PRIMARY OUTCOMES:
Reduction or discontinuation of the DMARD therapy in relation to the Covid-19 sanitary crisis | 1 Day
  Reduction or discontinuation of treatment with sDMARD, bDMARD or tsDMARD

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning one month and ending five years following the end study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.